CLINICAL TRIAL: NCT01708577
Title: Ultra High Speed Mobile Information and Communication
Brief Title: UMIC Validation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 11-111; EK 180/11 (Other: Ethics Committee University Hospital Aachen)
Record Dates: First submitted 2012-09-28; First posted 2012-10-17 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Healthy
Keywords: heart rate; sweating; respiration; acceleration of body movement; heart activity.
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IPANEMA validation without water intake (Experimental): The one group is restricted to the water intake during the Indoor phase during testing the IPANEMA measurement system. The other group is not restricted to the water intake.
  Interventions: Device: Validation of the IPANEMA - measurement system
- IPANEMA validation with water intake (Experimental): The one group is restricted to the water intake during the Indoor phase, the other group is not restricted to the water intake.
  Interventions: Device: Validation of the IPANEMA - measurement system

INTERVENTIONS:
Device: Validation of the IPANEMA - measurement system — Control of the body conditions under real life conditions during a sportive activity.

SUMMARY:
The purpose of the study is to evaluate the feasibility of a new wearable computerised system designed for an ongoing monitoring of sportsmen under real-life conditions. This system consists of different sensors and Bluetooth Transmitters interconnected by wires and integrated in the textile of a T-shirt. Several physiologic parameters including bioimpedance should be investigated under conditions relevant for an intensive physical activity, like high body temperature or partial dehydration. This system has to be tested under laboratory and "natural/open air" conditions, the obtained evaluations compared with standardised established diagnostic methods.

DETAILED DESCRIPTION:
The new wearable sensor- and monitoring system has to be tested on 20 healthy sportsmen of both genders in the age between 18 and 35 years. The aim of the present study is the characterisation of technical parameters, diagnostic precision and practical applicability of this system, which should be able to measure and translate information of actual physiologic state during the physical activity of sportsmen under real-life conditions.

IPANEMA (Integrated Posture and Activity Network) is a construct consisting of electrodes and several specialized sensors integrated in the textile tissue of a T-Shirt and interconnected with "electronic nods", an equipment supporting the central computerized control system with information via Bluetooth signals.

This body sensor network enables ablations of electrical activity of heart (ECG), Bioimpedance Spectroscopy (BIS), measuring of temperature and humidity on the surface of skin, breathing intensity and acceleration of body movement.

The study is divided in 3 parts, the indoor part, the outdoor part, and the part of measurements under controlled artificial temperature conditions (climate chamber).

The outdoor measurements will be performed at different running tracks, e.g. at the Hochschulsportzentrum, Lousberg, and can be separated in two subtypes, the training and the competition.

The indoor study phase lasts ca. 2 hours, where the volunteers will be analysed during running on a tread mill with both, the IPANEMA system and common medical monitoring procedures. The evaluations of identical physiological parameters obtained by use of stationary diagnostic equipment, the ergospirometric device PowerCube Ergo, BIS measurement system Xitron Hydra 4200, infra-red camera VarioCam®hr-basic and standard medical ECG measurements are used as reference values. Two hours before the start and during the entire training phase, the experimental group is restricted to food and liquid intake in opposite to control group. These experimental conditions purpose to clarify several physiological effects of dehydration during sportive activities. The outdoor- and climate chamber- investigations do not prescribe the liquid deprivation.

The climate chamber measurements will be performed in a temperature controlled room. This measurement session can last up to 3 hours and temperature inside of climate chamber can be increased until 40Cº. Such conditions may simulate body sensor network and elicit physiological effects comparable to effects obtained during sportive activities. No sport is performed by volunteers during the climate chamber phase.

ELIGIBILITY:
Inclusion Criteria:

* healthy, sporty person
* age 18-35 years
* able to give informed consent

Exclusion Criteria:

* electrophobics
* metallic and / or electric implants
* balance difficulties
* cardiac insufficiency
* arterial hypotension
* truncal ataxia
* underage persons
* pregnancy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-07; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Determination of vital signs out of a portable measuring system for monitoring performance of athletes during exercise | ten measurements each three hours
  Validation of a new portable und functional sensor based monitoring system.

SECONDARY OUTCOMES:
Determination of vital signs out of a new textile integrated and portable measurement system during training and competition conditions in comparision to parallel measurements with the reference devices | ten measurements each three hours
  Due to the design and type of measurements the study is divided into 3 parts, Indoor, Outdoor and Climate Chamber. The measurement duration for every part lasts 2-3 hours. The obtained data will be compared to results obtained by conventional methods. It includes the precision of measurement, the transfer of data and validation of computer supported data analysis. The measured parameters include temperature of the body, humidity on the body surface, ECG, volume and rate of breathing

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Krüger, Univ.-Prof., Principal Investigator — Internal Medicine I, University Hospital Aachen
Locations (1):
- Internal Medicine I, University Hospital, Aachen, North Rhine-Westphalia, Germany